CLINICAL TRIAL: NCT05395481
Title: A Single-Ascending and Repeated Subcutaneous Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3849891 in Participants With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) Who Have the PNPLA3 I148M Genotype
Brief Title: A Single-Ascending and Repeated Dose Study of LY3849891 in Participants With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18214; J3W-MC-GZOA (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Dysfunction-Associated Steatohepatitis (MASH); Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD)
Keywords: Hepatic fibrosis; Biomarkers; Magnetic resonance imaging; Pharmacokinetics; Liver fat
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3849891 (Part A) (Experimental): Single ascending doses of LY3849891 administered subcutaneously (SC)
  Interventions: Drug: LY3849891
- LY3849891 (Part B) (Experimental): Repeated doses of LY3849891 administered SC
  Interventions: Drug: LY3849891
- Placebo (Part A) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3849891 — Administered SC
  Arms: LY3849891 (Part A); LY3849891 (Part B)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug LY3849891 in participants with metabolic dysfunction-associated steatotic liver disease (MASLD) who have the patatin-like phospholipase domain-containing protein 3 (PNPLA3) I148M genotype. Blood tests and magnetic resonance imaging of the liver will be performed to determine the effects of LY3849891 on MASLD and assessment of resolution of liver fibroinflammation. Blood tests will also determine how long it takes the body to eliminate LY3849891. This is a 2-part study and may last up to 32 weeks for each participant and may include 12 visits in parts A and B.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (BMI) within the range greater than or equal to (≥) 25 and less than (<) 50 kilogram per square meter (kg/m²) inclusive
* Participants must have liver fat content ≥10% in Part A and ≥8% for Part B as determined by MRI-PDFF
* Participants must be carriers of the PNPLA3 I148M allele
* Participants with or without type 2 diabetes mellitus (T2DM)

  o For participants with T2DM, hemoglobin A1c (HbA1c) <8% in Part A and <9% in Part B
* Male participants agree to use an effective method of contraception for the duration of the study and for 90 days after the last dose of study intervention
* Women not of childbearing potential may participate and include those who are: infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as Mullerian agenesis; or those who are postmenopausal

Exclusion Criteria:

* Participants must not have known or suspected alcohol abuse (>14 units/week for women and >21 units/week for men) or active substance abuse
* Participants must not have evidence of cirrhosis or other forms of liver disease
* Participants must not have heart attack, stroke, or hospitalization for congestive heart failure in the past 3 months
* Participants must not have active cancer within the last 5 years
* Participants must not have uncontrolled high blood pressure
* Participants must not have renal impairment with estimated glomerular filtration rate (eGFR) <60 milliliter per minute per 1.73 square meter (ml/min/1.73m²)
* Participants must not have a diagnosis of type 1 diabetes
* Participants must not have a contraindication to MRI examinations, such as persons with cardiac pacemaker and implants made out of metal (for example, cochlear implant, nerve stimulators, magnetic vascular clips, and metallic heart valve) or other contraindications for MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Adverse Event(s) (AEs) Considered by the Investigator to be Related to Study Drug Administration | Predose up to 26 weeks post dose
  A summary of TEAEs and AEs, regardless of causality, will be reported in the Reported Adverse Events module
Part B: Pharmacodynamics (PD): Mean change from baseline on liver inflammation and fibrosis measured by magnetic resonance imaging (MRI) | Baseline through 24 weeks
  PD: Mean change from baseline on liver inflammation and fibrosis content measured by MRI

SECONDARY OUTCOMES:
Part A: PD: Liver fat content measured by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Predose through Week 26
  Part A: PD: Liver fat content measured by (MRI-PDFF)
Part A: PK: Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC(0-inf)) of LY3849891 | Predose through Week 26
  Part A: PK: AUC(0-inf) of LY3849891
Part A: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3849891 | Predose through Week 26
  Part A: PK: Cmax of LY3849891
Part A: PK: Time to Maximum Observed Concentration (Tmax) of LY3849891 | Predose through Week 26
  Part A: PK: Tmax of LY3849891
Part B: PD: Liver fat content changes at baseline and specified timepoints by MRI-PDFF | Predose through Week 24
  Part B: PD: Liver fat content changes at baseline and specified timepoints by MRI-PDFF
Part B: PK: AUC(0-inf) of LY3849891 and its Metabolite | Predose through Week 24
  Part B: PK: AUC(0-inf) of LY3849891 and its metabolite
Part B: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3849891 and its metabolite | Predose through Week 24
  Part B: PK: Cmax of LY3849891 and its metabolite
Part B: PK: Tmax of LY3849891 and its metabolite | Predose through Week 24
  Part B: PK: Tmax of LY3849891 and its metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- United States (13):
  - Arizona Liver Health - Chandler, Chandler, Arizona
  - Orange County Research Center, Orange, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Synergy Healthcare LLC, Brandon, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - Evolution Clinical Trials, Inc, Miami, Florida
  - Advanced Pharma Clinical Research, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - IU Health University Hospital, Indianapolis, Indiana
  - Houston Research Institute, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
- Japan (2):
  - P-One Clinic, Hachiōji
  - Clinical Research Hospital Tokyo, Shinjuku-ku
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Single-Ascending and Repeated Dose Study of LY3849891 in Participants With Nonalcoholic Fatty Liver Disease — https://trials.lillytrialguide.com/en-US/trial/7Mr5aA8joiUc52P5C9UXKa